CLINICAL TRIAL: NCT07186660
Title: Evaluation of a Novel Insulin Sensitizer on Glycemic Control, Insulin Usage, and Cardiovascular Biomarkers in People With Type 1 Diabetes Who Use Closed-loop Automated Insulin Delivery
Brief Title: Evaluation of a Novel Insulin Sensitizer in People With Type 1 Diabetes
Acronym: WBH003
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, William Horton, MD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 302645; 3-SRA-2025-1773-M-B (Other Grant/Funding Number: Breakthrough T1D)
Record Dates: First submitted 2025-09-12; First posted 2025-09-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes (T1D); Glycemic Control for Diabetes Mellitus; Insulin; Ketones; Cardiovascular Health
Keywords: Type 1 Diabetes; closed loop technology; time-in-range; adjunct therapy; cardiovascular health
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Ketosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinical research team
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CIR-0602K (Active Comparator): CIR-0602K 250 mg daily
  Interventions: Drug: CIR-0602K
- Placebo (Placebo Comparator): Matching Placebo Tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CIR-0602K — mitochondrial pyruvate carrier inhibitor
  Arms: CIR-0602K
Drug: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if the study drug CIR-0602K will improve glucose time-in-range and/or lower total daily insulin dose in people with type 1 diabetes who are using closed-loop automated insulin delivery. Researchers will compare CIR-0602K to a placebo (a look-alike substance that contains no drug) to see if it achieves the investigational endpoints. If the study results show that the drug works to increase time-in-range and lower insulin doses, this will lead to further studies which may then make the drug available to the public.

DETAILED DESCRIPTION:
Participants in the study will:

* Come to the Clinical Research Unit (CRU) at UVA Medical Center for 3 visits: Screening, Baseline (Admission 1) and End-of-Study (Admission 2).
* Complete various tests of cardiovascular health at each visit.
* Take either an experimental drug (CIR-0602K) or placebo for 12 weeks.
* Wear a study CGM with their personal insulin pump for 12 weeks.
* Be given a ketone meter and strips and be asked to take a fingerstick ketone reading every morning for 12 weeks.
* The study team will contact the participants regularly during the study to check their health and how they are tolerating the study drug/placebo.
* Return the study CGM, ketone meter, and remaining supplies, etc. at the end of the study.
* Notify the study team of any illness, injury, hypoglycemic or hyperglycemic events during the study

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. History of type 1 diabetes for at least one year
4. Age 18-45 years
5. HbA1c <10%

   * BMI 18-35 kg/m2. Within this criterion, participants must have either BMI ≥25 or total daily insulin dose of ≥0.5 units/kg/day.
   * Currently utilizing closed-loop AID therapy that is compatible with Dexcom G7 CGM.
   * On stable regimen of non-diabetic medications for the last 6 months.
   * All screening labs within normal limits or not clinically significant.
   * Ability to take oral medication and be willing to adhere to the study drug/placebo for 12 weeks.
   * For females and males of reproductive potential: agreement to use adequate contraception during study participation and for an additional 2 weeks after the end of CIR-0602K administration.
   * For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner during study intervention.
   * Agreement to adhere to Lifestyle Considerations throughout study duration.

Exclusion Criteria:

* Current Pregnancy or currently breastfeeding.
* History of smoking tobacco products within the last two years.
* History of alcohol abuse or illicit drug abuse within 6 months of screening.
* Known history of human immunodeficiency virus (HIV).
* History of other significant disease (e.g., cardiac, cerebrovascular, gastrointestinal, liver, renal, or endocrine) that could, in the investigator's view, alter study outcomes
* Any surgical or medical condition which may significantly alter the absorption of the study drug including but not limited to the following: history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling, or gastric banding, currently active inflammatory bowel syndrome.
* Current use of any antihyperglycemic medication beyond insulin (i.e., GLP-1 receptor agonists, SGLT2 inhibitors, etc.).
* Unstable doses (i.e., dose change within the last 4 months) of vasoactive medications (e.g., calcium-channel blockers, statins, angiotensin-converting enzyme inhibitors, diuretics, nitrates, alpha-blockers, beta-blockers, etc.).
* Daily use of anti-inflammatory medications (e.g., ibuprofen, aspirin, prednisone, dexamethasone, etc.).
* Diagnosis of peripheral neuropathy (assessed by screening monofilament exam).
* Macroalbuminuria (i.e., urine albumin: creatinine >300 mg per g).
* Retinopathy beyond mild, nonproliferative retinopathy.
* History of Level 3 hypoglycemia within the last 12 months.
* History of diabetic ketoacidosis (DKA) within the last 12 months.
* Screening electrocardiogram (ECG) findings indicative of arrhythmia, sinus node disease, or ischemic heart disease.
* Screening oxygen saturation <90%
* History of hypersensitivity or prior adverse reaction to the study drug, closely-related compounds, or any of the stated ingredients.
* Use of concomitant medications with a known significant metabolism by CYP2C8 or CYP2C (including paclitaxel, phenytoin, warfarin, celecoxib, tolbutamide, or repaglinide) for the duration of the study.
* Participation in an investigational study (other than a non-treatment registry study) or received an investigational drug withing 30 days or 5 half-lives (whichever is longer) prior to randomization.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Glucose Time-in-Range | 12 weeks
  Glucose time 70-180 mg/dL

SECONDARY OUTCOMES:
Total Daily Insulin Dose | 12 weeks
  Units of insulin per day
Glucose Time-above-Range | 12 weeks
  Glucose time >180 mg/dL
Glucose Time-Below-Range | 12 weeks
  Glucose time <70 mg/dL
Hemoglobin A1c | 12 weeks
  measure of glycemic control
Insulin Sensitivity | 12 weeks
  M-value from euglycemic insulin clamp

OTHER OUTCOMES:
Brachial Artery Flow-Mediated Dilation | 12 weeks
  Noninvasive measurement of blood vessel function
Carotid-Femoral Pulse Wave Velocity | 12 weeks
  Noninvasive measure of aortic stiffness
Radial Artery Augmentation Index | 12 weeks
  Noninvasive measure of radial artery stiffness
C-peptide | 12 weeks
  Blood test that measures endogenous insulin secretion
Daily fasting ketone level | 12 weeks
  Measure of blood ketone level collected by fingerstick meter conducted at home each morning
Cardiovascular Biomarkers | 12 weeks
  IL-6, TNF-alpha, hsCRP, E-selectin, ICAM-1, adiponectin
Peripheral Blood Mononuclear Cells | 12 weeks
  CD14++CD16-

CONTACTS AND LOCATIONS:
Overall Officials: William B. Horton, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigative team will finalize the decision (as to whether or not to share IPD) at a later date. Of note, IPD in this study qualifies as protected health information and would thus require safety considerations.